CLINICAL TRIAL: NCT05885386
Title: A Study on the Safety and Effectiveness of Temozolomide for Neoadjuvant Treatment of Pheochromocytoma or Paraganglioma Patients
Brief Title: A Study on the Safety and Effectiveness of Temozolomide for Neoadjuvant Treatment of PPGL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06086-05
Record Dates: First submitted 2023-05-22; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Pheochromocytoma; Paraganglioma
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma | interventions — Temozolomide

STUDY DESIGN:
Intervention Model Description: PPGLs could not be performed R0 resection due to the large tumor size and close relationship with surrounding tissues (blood vessels, kidneys, pancreas, liver, etc.)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pheochromocytoma or Paraganglioma patients (Other): TMZ was administered orally at an initial daily dose of 150 mg/m2 per day for 5 days, every 28 days preoperatively. In patients with a good tolerance during the first cycle, the dose was increased to 200 mg/m2 per day for 5 days, every 28 days.
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide — TMZ was administered orally at an initial daily dose of 150 mg/m2 per day for 5 days, every 28 days preoperatively. In patients with a good tolerance during the first cycle, the dose was increased to 200 mg/m2 per day for 5 days, every 28 days.

SUMMARY:
This phase II trial studies the effectiveness oftemozolomide in the neoadjuvant therapy oflocally advanced,or unresectable pheochromocytoma or paragangliom(PPGL). Temozolomide (TMZ) is a novel oral alkylation chemotherapeutic agent. Inthisstudy,temozolomidewill be used preoperatively in order to change unresectable tumors to resectable and reduce the high risk of surgery.

DETAILED DESCRIPTION:
The first choice for the treatment of PPGL is surgery. PPGL can be cured by complete resection of the lesion. However, some PPGLs could not be performed R0 resection due to the large tumor size and close relationship with surrounding tissues (blood vessels, kidneys, pancreas, liver, etc.). In this case, in order to achieve R0 resection, they need to undergo expand the scope of surgery, such as simultaneous resection of vital organs,and with extreamly high risks.There is no treatment option for those locally advanced or unresectable PPGLpatients currently. Temozolomide (TMZ), an oral alkylation chemotherapeutic agent, has been used in recent years and shown to have beneficial effects on metastatic PPGL with few side effects. TMZ has been recommended in National Comprehensive Cancer Network (NCCN) Guidelines Version 1.2022 for treating metastatic PPGL patients. This prospective, single arm, phase II study is designed to evaluate the efficacy of neoadjuvant therapy with TMZ in locally advanced,or unresectable PPGL patients or patients with severe catecholamine cardiomyopathy who are intolerance of operation.TMZ was administered orally at an initial daily dose of 150 mg/m2 per day for 5 days, every 28 days preoperatively. In patients with a good tolerance during the first cycle, the dose was increased to 200 mg/m2 per day for 5 days, every 28 days. Imaging examinations will be conducted after3 courses to re-evaluate the surgical possibility and surgery risks. If the patient's tumor shrinks after 3 courses but is still unresectable, the patients will continue TMZ therapy for another 3 courses.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent.
* Age 10-70 years old
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2.
* The patient is diagnosed as pheochromocytoma or paraganglioma which is unresectable with R0 surgery, or extensive and thus maybe requiring resection of important organs, or Inoperable due to heart and other complications, or with very high surgical risk.
* Estimated life expectancy longer than 6 months.
* Confirmed non-pregnancy and lactation. During the entire study period and within 6 months after the last administration, the subjects and their spouses are willing to use efficient contraceptive measures.
* Laboratory requirements:

  * Absolute granulocyte count (AGC) greater than 1.5 x 109/L;
  * Platelet count greater than 80 x 109/L; 3) Hemoglobin greater than 90g/L;
  * Serum bilirubin less than 1.5 x upper limit of normal (ULN);
  * Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 2.5 x ULN; Serum creatinine less than 1.5 x ULN or creatinine clearance (CCr)≥60ml/min;
  * Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ lower limit of normal value (50%).

Exclusion Criteria:

* Have other tumors.
* Patients were treated with other antitumor agents.
* Pregnant or nursing women.
* A history of allergic reactions to temozolomide or dacarbazine.
* Severe myelosuppression or abnormal coagulation.
* Severe liver and kidney insufficiency.
* Bowel obstruction or other conditions that interfere with taking medication.

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients whose tumor change from unresectable to resectable tumor | At the end of Cycle 3 (each cycle is 28 days)
  The proportion of PPGL patients whose tumor change from unresectable to resectable

SECONDARY OUTCOMES:
the objective response rate (ORR) | At the end of Cycle 3 (each cycle is 28 days)
  Defined for all patients whose tumor met the criteria of Complete Response (CR)and Partial Response (PR)
The ratio of tumor shrinkage. | At the end of Cycle 3 (each cycle is 28 days)
  The proportion of decrease in the sum of total size of the target lesions after treatment compared to before treatment.
The biochemical response. | At the end of Cycle 3 (each cycle is 28 days)
  An effective response of 24hCA, MNs meant that the concentration decreaseed by more than 40% than the baseline value or decreaseed to the normal range.
R0 resection rate | At the end of Cycle 3 (each cycle is 28 days)
  The proportion of patients with surgical resection reached R0 resection
Major pathological response rate (MPR) | At the end of Cycle 3 (each cycle is 28 days)
  Defined as the remaining surviving tumor after surgical resection do not exceed 10% of the initial tumor tissue.
Pathologic complete remission (pCR) | At the end of Cycle 3 (each cycle is 28 days)
  There is no tumor cells microscopically.
Safety of temozolomide treatment | At the end of Cycle 1 (each cycle is 28 days)
  Incidence of adverse events assessed by Common Terminology Criteria for Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Anli Tong, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No